CLINICAL TRIAL: NCT00600704
Title: Impact of Fluid Restriction Policy Added to Intra-Operative Cell Salvage in Reducing the Use of Red Cells in Cardiac Surgery
Brief Title: Impact of Fluid Restriction Policy in Reducing the Use of Red Cells in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: ATHINA KLEITSAKI, LARISSA UNIVERSITY HOSPITAL/DPT OF ANESTHESIOLOGY
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LUH 1975 AK; POL 1969 TT
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass; Erythrocyte Transfusion
Keywords: Allogenic Blood Use; Total Blood Loss; Reinfusion of Washed Shed Blood
MeSH Terms: conditions — Coronary Artery Disease; Exsanguination

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RESTRICTED FLUIDS (Active Comparator): Infusion of Hes 130/0.4 up to 500 ml until the beginning of Cardiopulmonary Bypass
  Interventions: Procedure: Fluid Restriction Policy
- FREE FLUIDS (Active Comparator): Free fluid infusion unless Hb< 6g/dl(allogenic blood use), until the beginning of Cardiopulmonary bypass
  Interventions: Procedure: Free fluid infusion

INTERVENTIONS:
Procedure: Fluid Restriction Policy — Infusion of Hes 130/0.4 up to 500 ml until the beginning of Cardiopulmonary bypass
  Arms: RESTRICTED FLUIDS
Procedure: Free fluid infusion — Free fluid infusion unless Hb< 6g/dl(allogenic blood use), until the beginning of Cardiopulmonary bypass
  Arms: FREE FLUIDS

SUMMARY:
The investigators' hypothesis is that restriction of circulating fluids in comparison to a liberal fluid administration policy would lead to a reduction of allogenic red blood cells exposure in patients undergoing cardiopulmonary bypass (CPB) for primary coronary artery bypass graft supported by reinfusion of washed shed blood from thoracic cavities.

DETAILED DESCRIPTION:
192 patients operated under equal conditions were assigned prospectively and randomly either for a restrictive protocol for intravenous fluid administration (group A, 100 patients) or not (group B, 92 patients). Transfusion guidelines were common for the two groups. The volumes of intravenous fluids, priming, "extra" volume on pump and cardioplegic solution and the volume of urine were recorded. Net erythrocyte volume loss was calculated. The number of the transfused PRC was analyzed as a continuous variable. "Transfusion" was analyzed as a categorical characteristic. Analysis employed Student's two-tailed t-test, t-paired test and chitest.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction (EF) of left ventricle (LV) > 35%
* Preoperative serum Creatinine < 150 μmol/l
* Preoperative Haemoglobin > 10/dl
* Peripheral anastomosis scheduled =< 3

Exclusion Criteria:

* redo bypass-emergency operations
* prior coronal stenting
* active congestive heart failure
* documented Myocardial Infraction within the previous 6 weeks
* NYHA class > 3
* Carotid stenosis > 50%
* CVA
* INR > 1.5
* chronic obstructive pulmonary disease (COPD)
* Steroid therapy-chronic inflammatory process
* Use of aprotinin or tranexamic acid

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ATHINA KLEITSAKI, Dr, Principal Investigator — Larissa University Hospital; GEORGE VRETZAKIS, M.D. PhD, Study Director — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; KONSTANTINOS STAMOULIS, M.D., Study Chair — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; CHRISTOS DRAGOUMANIS, M.D. PhD, Study Chair — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; VASILIOS TASOUDIS, M.D., Study Chair — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; KATERINA KYRIAKAKI, M.D., Study Chair — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; DEMETRIOS MIKROULIS, M.D. PhD, Study Chair — Department of Cardiothoracic Surgery, University Hospital of Larissa, Greece; ATHANASIOS GIANNOUKAS, MD MSc PhD, Study Chair — Department of Vascular Surgery, University Hospital of Larissa, Greece; NIKOLAOS TSILIMINGAS, M.D. PhD, Study Chair — Department of Cardiothoracic Surgery, University Hospital of Larissa, Greece
Locations (1):
- Larissa University Hospital, Larissa, Thesalia, Greece

REFERENCES:
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454
- [Background] Dial S, Delabays E, Albert M, Gonzalez A, Camarda J, Law A, Menzies D. Hemodilution and surgical hemostasis contribute significantly to transfusion requirements in patients undergoing coronary artery bypass. J Thorac Cardiovasc Surg. 2005 Sep;130(3):654-61. doi: 10.1016/j.jtcvs.2005.02.025. PMID 16153909
- [Background] Stover EP, Siegel LC, Parks R, Levin J, Body SC, Maddi R, D'Ambra MN, Mangano DT, Spiess BD. Variability in transfusion practice for coronary artery bypass surgery persists despite national consensus guidelines: a 24-institution study. Institutions of the Multicenter Study of Perioperative Ischemia Research Group. Anesthesiology. 1998 Feb;88(2):327-33. doi: 10.1097/00000542-199802000-00009. PMID 9477051
- [Background] Karkouti K, Djaiani G, Borger MA, Beattie WS, Fedorko L, Wijeysundera D, Ivanov J, Karski J. Low hematocrit during cardiopulmonary bypass is associated with increased risk of perioperative stroke in cardiac surgery. Ann Thorac Surg. 2005 Oct;80(4):1381-7. doi: 10.1016/j.athoracsur.2005.03.137. PMID 16181875
- [Background] Habib RH, Zacharias A, Schwann TA, Riordan CJ, Durham SJ, Shah A. Adverse effects of low hematocrit during cardiopulmonary bypass in the adult: should current practice be changed? J Thorac Cardiovasc Surg. 2003 Jun;125(6):1438-50. doi: 10.1016/s0022-5223(02)73291-1. PMID 12830066
- [Background] DeFoe GR, Ross CS, Olmstead EM, Surgenor SD, Fillinger MP, Groom RC, Forest RJ, Pieroni JW, Warren CS, Bogosian ME, Krumholz CF, Clark C, Clough RA, Weldner PW, Lahey SJ, Leavitt BJ, Marrin CA, Charlesworth DC, Marshall P, O'Connor GT. Lowest hematocrit on bypass and adverse outcomes associated with coronary artery bypass grafting. Northern New England Cardiovascular Disease Study Group. Ann Thorac Surg. 2001 Mar;71(3):769-76. doi: 10.1016/s0003-4975(00)02393-6. PMID 11269449
- [Derived] Vretzakis G, Kleitsaki A, Stamoulis K, Dragoumanis C, Tasoudis V, Kyriakaki K, Mikroulis D, Giannoukas A, Tsilimingas N. The impact of fluid restriction policy in reducing the use of red blood cells in cardiac surgery. Acta Anaesthesiol Belg. 2009;60(4):221-8. PMID 20187484
- [Derived] Vretzakis G, Kleitsaki A, Stamoulis K, Bareka M, Georgopoulou S, Karanikolas M, Giannoukas A. Intra-operative intravenous fluid restriction reduces perioperative red blood cell transfusion in elective cardiac surgery, especially in transfusion-prone patients: a prospective, randomized controlled trial. J Cardiothorac Surg. 2010 Feb 24;5:7. doi: 10.1186/1749-8090-5-7. PMID 20181257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective study was conducted in our University Hospital over a 20-month period, after approval from the Institution Ethics committee, and written informed consent was obtained from all patients before entering the study. All the participants were patients of the Cardio-Thoracic Clinic of our Hospital.
Pre-assignment Details: Exclusion criteria were emergency or re-do operations, operations starting after 18.00, administration of tissue plasminogen activator (TPA) or other thrombolytic medications, pre-existing hematologic disease or coagulation abnormality, advanced cirrhosis, renal failure, preoperative blood product transfusion, combined cardiac and carotid surgery.
Groups:
- RESTRICTED FLUIDS: Infusion of Hes 130/0.4 up to 500 ml
- FREE FLUIDS: Free fluid infusion unless Hb< 6g/dl(allogenic blood use)
Period: Overall Study
Arm/Group | RESTRICTED FLUIDS | FREE FLUIDS
Started | 100 | 92
Completed | 100 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RESTRICTED FLUIDS | FREE FLUIDS | Total
Number analyzed (Participants) | 100 | 92 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 92 | 192
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (7.9) | 65.5 (8.3) | 65.77 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 83 | 76 | 159
Region of Enrollment [Number; unit: participants]
  Greece | 100 | 92 | 192

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Packed Red Cells Units Transfused During Hospital Stay
Time Frame: 20 months
Population: Patients between ages 18-85 undergoing elective cardiac surgery under cardiopulmonary bypass
Measure: Mean (95% Confidence Interval); unit: packed red cells units
Units Other Than Participants: PRC Units
Arm/Group | RESTRICTED FLUIDS | FREE FLUIDS
Number analyzed (Participants) | 100 | 92
Number analyzed (PRC Units) | 113 | 176
packed red cells units | 1.13 [0.90 to 1.36] | 1.91 [1.63 to 2.19]
Statistical Analysis 1: Comparison: RESTRICTED FLUIDS vs FREE FLUIDS; Sample size calculation was based on a two-sided alpha error of .05 and 80% power. After applying the protocol in two equal groups of 10 patients, the analysis showed that the study requires 60 patients per group. However, we decided to enroll up to 100 patients per group to allow for patient attrition or missing data, and also in order to look for differences with regards to transfusion between patient subgroups; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.379, 95% CI 2-sided [0.189 to 0.569], Standard Deviation 0.096
Statistical Analysis 2: Comparison: RESTRICTED FLUIDS vs FREE FLUIDS; Null hypothesis :restrictive fluid protocol does not have any effect concerning the mean number of PRC units transfused; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.797, 95% CI 2-sided [0.465 to 1.129], Standard Error of Mean 0.168 — The mean difference between groups B and A is adjusted for age, gender, BMI and preoperative HCT, while BSA, weight, height, postoperative HCT were not included in the final model to avoid collinearity

ADVERSE EVENTS:
Arm/Group | RESTRICTED FLUIDS | FREE FLUIDS
Serious Adverse Events (participants affected / at risk) | 20/100 | 18/92
Other Adverse Events (participants affected / at risk) | 2/100 | 2/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RESTRICTED FLUIDS (N=100) | FREE FLUIDS (N=92)
myocardial infraction (Cardiac disorders) | 5 (5) | 4 (4)
persistent significant arrythmia (Cardiac disorders) | 8 (8) | 6 (6)
low output syndrome (Congenital, familial and genetic disorders) | 6 (6) | 7 (7)
persistent neurological dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
lower extremity ischemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RESTRICTED FLUIDS (N=100) | FREE FLUIDS (N=92)
reoperation for bleeding (Surgical and medical procedures) | 1/1 (1) | 1/1 (1)
renal failure (Renal and urinary disorders) | 1/1 (1) | 1/1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes